CLINICAL TRIAL: NCT02403024
Title: I-Walk-CRC - Feasibility and Efficacy of Interval Walking in Patients With Colorectal Cancer
Brief Title: Feasibility and Efficacy of Interval Walking in Patients With Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Jesper Frank Christensen, PhD, Post doc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I-Walk-CRC
Record Dates: First submitted 2015-03-24; First posted 2015-03-31 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Colorectal Cancer
Keywords: Colon cancer; rectal cancer; exercise; physical activity; metabolic health
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- InterWalk (Experimental): The intervention program will prescribe that patients performing 150 min of interval training per week.
  Interventions: Behavioral: InterWalk
- Waiting list Control (Other): Patients allocated to the waiting-list control group will receive usual care control for the first 12 weeks of the study and will receive the same instructions for download and use of the InterWalk app in the final 12 weeks.
  Interventions: Behavioral: Waiting list control

INTERVENTIONS:
Behavioral: InterWalk — Patient allocated to the InterWalk-group will be introduced to the InterWalk app, including instructions on how to down load and use the application. and prescribed to perform Interval Walking for 150 min per week
  Arms: InterWalk
Behavioral: Waiting list control — Patients allocated to the waiting-list control group will be prescribed standard guidelines for the patient group, but will be asked not to download and use the InterWalk app (which is freely available) for the first 12 weeks of the study period. After the first 12 weeks (the control period), patients in this group will receive the same instructions for download and use of the InterWalk app in the following 12 weeks
  Arms: Waiting list Control

SUMMARY:
Background: The level physical exercise is strongly associated with colorectal cancer risk in the general population, and recent data shows that physical activity after a colorectal cancer diagnosis is inversely associated with mortality risk, indication the physical exercise can protect against disease progression. However, few studies have successfully performed exercise interventions in patients with colorectal cancer, and the potential mechanisms responsible for the tumor suppressing effects of exercise remain poorly explored.

Purpose: To investigate interval-walking, delivered by the InterWalk smart phone application as exercise-modality in patients with colorectal cancer. Specifically it is the aim to explore if InterWalk is safe and feasible as well as effective to improve cardio-metabolic health profile.

Subjects: Colorectal cancer patients, stage I-III, who are at least one month post-surgery and have concluded any adjuvant chemotherapy treatment, are eligible for inclusion. Exclusion criteria are: age <18; any major surgical procedure planned within 6 months after inclusion; pregnancy; ongoing treatment for any known malignancy; performance status > 1; unable to read and understand Danish

Methods: 40 colorectal cancer patients are included and randomized to I) InterWalk or II) waiting list control for 24 weeks. Patients are evaluated at baseline, week 12 and week 24 by assessment measures to determine cardio-metabolic health profile and other relevant study outcomes, including: cardiopulmonary exercise test (VO2peak); anthropometrics; blood pressure; resting heart rate; body composition; health related quality of life questionnaires; plasma concentration levels of cholesterol, triglycerides, insulin, glucose and inflammatory cytokines; insulin sensitivity; and cognitive function.

DETAILED DESCRIPTION:
INTRODUCTION More than 30.000 individuals are living with a colorectal cancer (CRC) diagnosis in Denmark today. Due to marked advances in surgical and medical treatment, as well as novel screening programs, this number is expected to increase over the coming years. Numerous studies have shown that physical activity is inversely associated with colorectal cancer risk. A meta-analysis of 52 studies found that regular participation in physical activity reduced disease risk by 24% (HR: 0.76 , 95%Confidence Interval [95%CI]: 0.72 - 0.81). Recent evidence furthermore shows that physical activity after a CRC diagnosis is a strong independent predictor for overall survival, CRC-specific survival, and survival after disease relapse. CRC patients who adhere to the current recommendation of at least 150 min moderate intensity physical activity per week have an estimated 10-40% lower CRC-specific and 20-50% lower overall mortality risk in comparison to sedentary counterparts. The causative mechanisms responsible for this protective effect are not fully elucidated, but several studies have shown that metabolic health factors, i.e. overweight/adiposity, systemic levels of glucose, insulin, Insulin-like Growth Factor (IGF)-1, leptin, adiponectin and inflammatory cytokines (TNF-α, CRP) are associated with CRC prognosis. These factors are, under normal circumstances modifiable through physical activity and exercise, which may constitute a plausible mode of action, through which, exercise may reduce risk of disease progression as well as development and/or progression of cardio-metabolic co-morbid disorders.

BACKGROUND Over the last decade, more than 70 studies have explored the capacity of physical exercise to improve physiological (fitness, muscle strength, body composition) and psychosocial (fatigue, depression, emotional well-being) outcomes in patients with cancer during and after anti-neoplastic therapy and although CRC is among the most prevalent malignancies, few exercise-trials have been performed in this patient group. The reason for this notable low number of studies, relative to other common cancers in particular breast and prostate cancer, may be a number of disease and treatment specific phenomena, e.g. high prevalence of co-morbidities, stoma, late-effects from surgery or adjuvants therapies etc., which may complicate participation in traditional hospital-based exercise-programs, which is often comprised of fitness- and strength-training. A recent meta-analysis included just 3 randomized trials investigating exercise in CRC patients, and found positive effects exercise vs control on cardiovascular fitness; standardized mean difference: 0.59 [95%CI 0.25-0.93], P<0.01. A recent pilot study furthermore showed that home-based exercise improved several metabolic factors including reduction in body weight, plasma insulin levels and improved insulin sensitivity. Thus, these data indicate that CRC patients can improve cardio-metabolic health profile by physical exercise; however, the present body of research have included a total of less than 200 patients; explored various exercise-modalities, and applied inconsistent and/or indirect assessment-methods. To this end, there is a remaining need for high quality evidence describing effective exercise-interventions in CRC patients, particularly interventions aimed to be successfully implemented in clinical practice in case of positive results.

Interval training, as characterized by inter-changing cycles of high and low intensity exercise, have long been recognized as the most effective exercise-modality to improve cardiopulmonary fitness, and can furthermore induce equal or greater metabolic effects than continuous exercise over longer duration. Considerable challenges exists however, when performing high intensity interval exercise-training in clinical settings. This type of exercise often needs to be performed on ergometer bicycles or treadmills and organized as supervised, hospital-based training to ensure proper monitoring and feedback to participants for optimal exercise intensity and progression, which limits the dissemination potential beyond the trial period.

Center for Physical Activity Research (CFAS) have performed a number of trials showing that interval training can be performed as free-living interval-walking, consisting of repeating cycles of 3 minutes fast walking followed by 3 minutes slow walking with significant positive effects in cardio-metabolic health profile. Our studies show, that 16 weeks of interval-walking improved VO2peak (+4ml /kg/min) reduced bodyweight (-4 kg) and fat mass (-3 kg) in patients with type 2 diabetes. Moreover, interval-walking improved plasma lipid-profile, glucose metabolism and insulin sensitivity, in contrast to continuous walking, which was matched for training-volume and energy expenditure. In parallel with these intervention-studies, a smart-phone application, called InterWalk (www.InterWalk.dk), has been developed, which can deliver this training program of repeating cycles: 3 minutes fast walking followed by 3 minutes slow walking. The exercise-program is based on an individualized test-function with live-feedback, ensuring proper exercise-intensities (walking-speed), and can simultaneously store test- and training data (exercise-time, walking-speed, distance etc.) to an external server for research purposes. Preliminary data shows that three months home-based interval-walking using the InterWalk-application can improve fitness by ~10%. Thus, our preliminary data shows InterWalk can deliver an un-supervised, yet individualized, structured and objectively monitored exercise-program which can effectively improve cardio-metabolic health, and may be more applicable and feasible, compared to traditional hospital-based programs in stigmatized patient groups with major co-morbid complications.

The investigators therefore propose this intervention can have a great health promoting potential in patients with CRC; however previous work have found considerable barriers and complications associated with successful participation in exercise-programs for this patient group. Thus, the investigators intend to explore whether interval-walking, delivered by the InterWalk-app, is safe and feasible, and furthermore the investigatorsintend to explore if the intervention can cause similar positive effects as the investigators have seen previously in other clinical populations.

PURPOSE AND HYPOTHESES Based on promising results from studies in type 2 diabetes, it is the primary purpose of this study to investigate interval-walking via InterWalk-app as health promoting exercise-intervention in patients with CRC. Specifically it is the aim of this pilot study to determine the safety, feasibility, adherence and compliance of InterWalk; as well as evaluating effects on cardio-metabolic health profile, compared to a waiting-list control group.

RESEARCH PLAN This is a prospective, randomized controlled pilot-study in 40 CRC patients. The study is a collaboration between Center for Physical Activity Research, Rigshospitalet, Institut for Folkesundhedsvidenskab, Copenhagen University, Oncology Clinic, Rigshospitalet, Abdominalcenter K, Bispebjerg Hospital, Gastroenheden Hvidovre Hospital, and Patientforeningen for Tarmkræft.

Recruitment and Randomization CRC patients will be recruited from the oncology clinic, Rigshospitalet and the gastro-intestinal surgical ward at Hvidovre Hospital. Patients, who have undergone adjuvant chemotherapy, will be informed of the study during their final visit at the oncology clinic. Patients in active surveillance will be informed of the study at the first clinical visit, at least one month after surgery. The responsible clinicians and nurses in the clinical department will present patients with the written information of the study and gather contact information for interested participants to the study coordinator for more information of the study. Before any study related test-procedures are initiated, patients will sign informed consent, and undergo medical screening including former and present medication, physical examination including resting EKG by a study physician to determine if the patient can be included in the trial and subsequently scheduled for baseline assessment.

Following baseline-assessment patients will be allocated to one of two experimental arms I) InterWalk or II) waiting-list control. To account for potential bias, patients will be stratified by prior treatment (adjuvant chemotherapy/no adjuvant chemotherapy), which may have significant impact on study outcomes. A random allocation sequence of treatment assignments for each stratification group will be created by the trial biostatistician and concealed from the study personal. The study coordinator will inform the patient of the treatment assignment and the patient will remain in this group for the full study period.

Study Outcomes and Procedures

The test procedures involve a number of assessments which will be conducted 3 times during the study; at baseline, week 12 and week 24:

1. Body composition by DXA scan
2. Fasting blood sample for analyses of plasma biochemistry (cholesterol, triglycerides, inflammatory markers, HbA1C)
3. Oral Glucose Tolerance Test (OGTT) with repeated measures of plasma glucose, insulin and c-peptide
4. Health related Quality of Life questionnaires
5. Cognitive function
6. Cardio Pulmonary Exercise Test (VO2peak)

Statistical Considerations The primary analysis will compare difference in changes in study outcomes from 0 to 12 weeks between the two treatment arms InterWalk vs control. For the primary outcome, VO2peak, assuming a standard deviation of 2 ml/kg/min, 16 patients in each group will provide 80% power to detect a between group difference of +2 ml/kg/min in. To account for a potential attrition-rate of up to 20%, 20 patients will be included in each group.

The primary analysis is performed as a random effect model using study outcomes as dependent variables, the covariates "group", "time" and their interaction as fixed effects, and a random effect of "patient".

Dropouts and Missing Observations Patients who wish to drop-out of the study during the intervention-periods will be offered to remain in the study with regard to test-assessments. All analyses are performed as 'intention-to-treat' analyses, thus all patients will remain in the originally allocated treatment arms regardless of compliance to the intervention. Potential drop-outs and missing observations are handled by the "missing at random" principle.

Ethical Considerations This study, as described, is expected to include limited risks, adverse effects and discomfort for subjects. During all assessment procedures, a medical doctor will be present in case of discomfort or other medical problems. Should patients report discomfort or adverse reactions during interval-walking, the study coordinator in collaboration with the responsible clinicians, will determine if the programs needs to be adapted or terminated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a verified stage I-III CRC diagnosis who has
* All surgical and oncological treatments must be terminated

Exclusion Criteria:

* Any major surgical procedure planned within 6 months after inclusion
* Pregnancy
* Ongoing treatment for any known current malignancy
* Performance status > 1
* Inability to read and understand Danish
* Physically active for more than 150 minutes (moderate intensity) per week thus adhering to the current recommendations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-08; Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Change in VO2peak | Baseline to week 12
  On a stationary bicycle, the participants perform 3 minutes warm up on 70 Watt followed by a step-by-step incremental test with workload increasing by 20 Watt every minute until exhaustion with direct measurement of oxygen uptake and carbon dioxide excretion with gas-exchange online-measurement equipment (Cosmed Quark, Rome, Italy).

SECONDARY OUTCOMES:
Change in Body composition | Baseline-to-week 12; baseline-to-week 24; week 12-to-week 24
  Body weight and anthropometrics (height, waist and hip circumference) will be assessed using standard procedures. Resting heart rate and blood pressure (Microlife, BPA100) will be determined in a supine position. Body composition (fat mass, bone mass and fat-free mass) and bone mineral density are analyzed by whole-body dual-energy X-ray absorptiometry (DXA) scan (Lunar, Lunar Corporation Madison, Wisconsin, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body. Since the different chemical compounds in the body absorb the intensity of the X-rays differently, the scan allows for a valid determination of bone mass, fat mass and fat-free/bone-free mass
Changes in bloodbiochemistry from fasting blood samples | Baseline-to-week 12; baseline-to-week 24; week 12-to-week 24
  Patients will have a fasting blood (30ml EDTA) sample taken to determine fasting concentrations of cholesterol, triglycerides, inflammatory markers; HbA1C, leptin, adiponectin.
Changes in patient-reported Quality of Life | Baseline-to-week 12; baseline-to-week 24; week 12-to-week 24
  Patient reported outcomes include: Functional Assessment of Cancer Treatment (FACT)-C, International Physical Activity Questionnaires (I-PAQ), Pittsburgh Sleep Quality Index (PSQI) and Behavioral Exercise Regulations Questionnaire (BREC)-2.
Changes in insulin sensityvity by measure of Oral Glucose Tolerance Test (OGTT) | Baseline-to-week 12; baseline-to-week 24; week 12-to-week 24
  The patients undergo standard OGTT assessment, by drinking 75 g glucose mixed in 300 ml water and have 10 ml blood samples taken after 60 and 120 min for analyses of plasma glucose, insulin and C-peptide.
Change in VO2peak (secondary comparisons) | baseline-to-week24, week 12-to-week 24
  On a motorized treadmill, patients will perform a 5 min warm-up period on a walking speed corresponding to ~50% of the age-predicted HR-max. After a 3 min rest, the patients will perform a graded, walking VO2-peak with incremental inclination and speed every other minute (Technogym Runrace, Gambettola, Italy), using indirect calorimetry (CPET, Quark, Rom, Italy).

CONTACTS AND LOCATIONS:
Overall Officials: Jesper F Christensen, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Hvidovre Hospital, Hvidovre

REFERENCES:
- [Derived] Christensen JF, Sundberg A, Osterkamp J, Thorsen-Streit S, Nielsen AB, Olsen CK, Djurhuus SS, Simonsen C, Schauer T, Ellingsgaard H, Osterlind K, Krarup PM, Mosgaard C, Vistisen K, Tolver A, Pedersen BK, Hojman P. Interval Walking Improves Glycemic Control and Body Composition After Cancer Treatment: A Randomized Controlled Trial. J Clin Endocrinol Metab. 2019 Sep 1;104(9):3701-3712. doi: 10.1210/jc.2019-00590. PMID 31220283